CLINICAL TRIAL: NCT04989062
Title: Predicting Obesity Consequences Using Body Measure and Urine Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Li-Wen Lee, Consultant Radiologist, Chang Gung Memorial Hospital
Other Study IDs: 201901889A3
Record Dates: First submitted 2021-07-11; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Body Composition; Electric Impedance
Keywords: Non-Alcoholic Fatty Liver Disease; Body Composition; Electric Impedance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy children: Apparently healthy children at Year 1 to Year 6 in the primary school in Taiwan. Exclusion criteria are children with metal implant or splint, pacemaker implantation, limb defect or injury and pregnant.
  Interventions: Diagnostic Test: Fibroscan; Diagnostic Test: Bioelectrical impedance analysis; Diagnostic Test: Urine unclear magnetic resonance metabolomics; Diagnostic Test: Hand grip strength

INTERVENTIONS:
Diagnostic Test: Fibroscan — Controlled attenuation parameter and liver stiffness measurement are measured.
Diagnostic Test: Bioelectrical impedance analysis — Body composition measures including fat mass, fat-free mass, percentage body fat in total body and body segments are obtained.
Diagnostic Test: Urine unclear magnetic resonance metabolomics — Metabolites in the urine are estimated by 600 MHz nuclear magnetic resonance.
Diagnostic Test: Hand grip strength — Hand grip strength in both hands is measured by hand-held dynamometer.

SUMMARY:
This is a prospective observational study which will recruit up to 1200 participants over a two-year period to investigate whether non-invasive methods such as bioelectrical impedance analysis parameters and urine metabolic profile are predictors for pediatric non-alcoholic liver disease.

DETAILED DESCRIPTION:
Obesity is associated with non-alcoholic fatty liver in children. Currently, body mass index is used for stratification risk for non-alcoholic fatty liver disease in children. However, body mass index represents the adjusted weight status for height and may not be a perfect surrogate for body fatness. This study assumes that a combination of body measures including parameters of bioelectrical impedance analysis and hand grip strength may better represented body fatness and healthy status than body mass index. Moreover, non-alcoholic fatty liver disease is strongly associated with the metabolic syndrome and non-invasive urine metabolic profile may be used to predict the disease status. The aim of this study will be to develop non-invasive methods using body measures and urine metabolic profile to predict pediatric fatty liver disease.

This study will recruit 1200 apparently healthy children at Year 1 to Year 6 in the primary schools in Taiwan within a two-year period. A series of tests including body measures, bioelectrical impedance analysis, hand grip strength and urine metabolomics by nuclear magnetic resonance will be performed in each participant. These data will be used as features to predict the results of Fibroscan test.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy male or female children
* Students in Year 1 to Year 6 of primary schools

Exclusion Criteria:

* Unknown liver disease
* Metal implant or splint
* Pacemaker implantation
* Limb defect or injury
* Pregnancy

Ages: 6 Years to 13 Years | Sex: All
Age Groups: Child
Study Population: Participants in the Year 1 to Year 6 of primary school (aged 6-13 years) without liver disease will be recruited for body measure, urine sampling and Fibroscan test.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between bioelectrical impedance analysis parameters and the degree of fatty liver | 24 months
  Correlation body composition parameters by bioelectrical impedance analysis and controlled attenuation parameter by Fibroscan

SECONDARY OUTCOMES:
Correlation between urine metabolites and the degree of fatty liver | 24 months
  Correlation between urine metabolites by nuclear magnetic resonance and controlled attenuation value parameter by Fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wen Lee, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital, Chiayi, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No